CLINICAL TRIAL: NCT04587895
Title: Feasibility Study of an Individualized Exergame Training for Older Adults With Mobility Impairment and/or Urinary Incontinence
Brief Title: Feasibility Study of an Individualized Exergame Training for Older Adults With MI and/or UI (VITAAL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eling DeBruin (Other)
Responsible Party: Sponsor-Investigator, Eling DeBruin, Prof. Dr., Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BASEC-Nr.: 2020-00578
Record Dates: First submitted 2020-09-24; First posted 2020-10-14 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Urinary Incontinence; Mobility Impairment; Older Adults
Keywords: exergame; healthy ageing; feasibility
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MI Intervention (Experimental): The VITAAL exergame intervention for MI includes 36 training sessions with three sessions per week, each lasting around 45 minutes (30 minutes real training time) resulting in 12 weeks of training (two weeks of break/holiday allowed). A training session includes an individually calculated amount of strength, cognitive-motor and balance training, which remains the same over the 12 week intervention period.
  Interventions: Behavioral: VITAAL Exergame
- MI Control (Active Comparator): Participants of the MI control group are instructed to do a non-individualized conventional training including 15 minutes walking exercise (in nature or on treadmill) and additional 15 minutes of strength, balance, and cognitive-motor exercises (at the therapy centre or at home). The exercises are based on recommendations from the "Beratungsstelle für Unfallverhütung" (bfu). The participants will receive a training booklet with the exercises. In total there are three different training programs which are divided according to their level of difficulty. Participants are instructed to start with the first level for four weeks and then go on to the next level for another 4 weeks. The control group training in this study includes 36 training session with three sessions per week, each lasting around 45 minutes resulting in 12 weeks of training (two weeks of break/holiday allowed).
  Interventions: Behavioral: Conventional Training MI
- UI Intervention (Experimental): For the incontinent women in this study, the VITAAL exergame intervention will last over 12 weeks and consists of three parts 1) VITAAL exergame (2 sessions/week) lasting 45 minutes each (30 minutes real training time) at the physio centre, 2) PFM exercises according to a training booklet (3 sessions/week) lasting 10 minutes each at home and 3) education related to UI at home.
  Interventions: Behavioral: VITAAL Exergame
- UI Control (Active Comparator): The control group training will last over 12 weeks. The training sessions will be divided in three parts 1) 30 minutes of brisk walking (2 sessions/week, 2) PFM exercises according to a training booklet (3 sessions/week) lasting 10 minutes each at home and 3) education related to UI at home. The PFM training booklet will be based on two studies that showed a reduction of incontinence in older adults while performing group pelvic floor muscle training (PFMT) and mobility exercises. The PFMT program will consist of 4 PFM exercises and will be divided into three phases allowing for the gradual progression in treatment (from first to third month), with gradual increase in difficult exercises in terms of duration, repetition and position. Each phase will last four weeks.
  Interventions: Behavioral: Conventional Training UI

INTERVENTIONS:
Behavioral: VITAAL Exergame — 12 weeks training with the VITAAL Exergame. The VITAAL exergame is an individualized multicomponent exergame training based mostly on the prevention and slowing of physical and cognitive decline and its consequences. It mainly consists of three (four with UI) components; strength training, balance training, cognitive training and pelvic floor muscle training (PFMT) when suffering from UI.
  Arms: MI Intervention; UI Intervention
Behavioral: Conventional Training UI — 12 weeks non-individualized conventional training with a training booklet and additional walking exercise. The PFM training booklet is based on exercises that showed a reduction of incontinence in older adults while performing group pelvic floor muscle training (PFMT) and mobility exercises.
  Arms: UI Control
Behavioral: Conventional Training MI — 12 weeks non-individualized conventional training with a training booklet and additional walking exercise. The exercises are based on recommendations from the "Beratungsstelle für Unfallverhütung" (bfu).
  Arms: MI Control

SUMMARY:
This study examines the feasibility of an individualized video game training (VITAAL Exergame) for older adults with mobility impairments and/or urinary incontinence. In addition, the effect of the newly developed training program on motor and cognitive functions is examined. This study is a national study. The development of the exergame was carried out at the Fraunhofer AICOS research center in Portugal and further studies are being conducted in international collaboration with the University of Montréal in Canada, KU Leuven in Belgium and ETH Zurich. The Exergame consists of a video game based training, which is performed with step movements. These movements are detected by two sensors on the feet. The video game should make the training fun and motivate to train. The training will include specific cognitive and physical functions. Special emphasis will be put on a continuous interaction and integration of motor and cognitive functions. An intact cognitive-motor interaction as well as balance and strength form the basis for all everyday performances, especially for safe and accident-free movement in older adults. In the Exergame VITAAL, balance is trained with step-based games. Strength, especially leg strength, is trained through Tai-Chi-like movements/exercises.

The pelvic floor training takes place using a vaginal probe that measures the contractions of the pelvic floor. The training games on the VITAAL Exergame have been adapted for this purpose and are controlled via the probe.

All participants receive an individually tailored training session that is optimally adapted to their needs based on the results of the pre-measurement. Participants with urinary incontinence also receive an integrated pelvic floor training. The study includes 32-52 seniors with mobility impairments and 8-28 older adults with urinary incontinence. Balance and strength, gait pattern, cognitive functions and pelvic floor specific functions will be measured before and after the training in order to detect any changes. The training should be carried out during 12 weeks, with a maximum of two weeks break/holidays. There are two measurement dates with all examinations, whereby one measurement date lasts approx. 1.5 hours. All study participants can continue their everyday life as usual.

DETAILED DESCRIPTION:
The VITAAL exergame is an individualized multicomponent exergame training based mostly on the prevention and slowing of physical and cognitive decline and its consequences. It mainly consists of three (four with UI) components; strength training, balance training, cognitive training and pelvic floor muscle training (PFMT) when suffering from UI. For strength training, Tai Chi-inspired movements are included which are a combination of classical strength exercises and Tai Chi movements. Since Tai Chi is mainly performed in a semi-squat posture it places a large load on the muscles of the lower extremities. For balance training, step-based training is included in the VITAAL exergame, as the execution of rapid and well directed steps has been shown to be effective in preventing falls. Both, Tai Chi-inspired exercises and step-based exercises, combined with challenging game tasks, provide a 'holistic' physical activity requiring motor functions, cognition and mental involvement. The PFMT is divided in two categories, isolated exercises of PFM (different contraction sequences) and dual task exercises, where PFM contractions are performed with or in combination with balance exercises. Moreover, Tai Chi-inspired training, step-based training and PFMT could be more motivating and joyful than standard exercises. Some cognitive training is already included in these training components as they represent simultaneous cognitive-motor interaction and require motor and cognitive functions. But specific attentional and executive functions are important for walking abilities and safe gait. Therefore, the VITAAL exergame explicitly targets on these neuropsychological functions (selective attention, divided attention, inhibition/interference control, mental flexibility, working memory). To maximize benefits for participants, the VITAAL exergame implements some basic general training principles; providing feedback, optimal load of task demands, progression of difficulty and high variability.

Intervention group MI:

The VITAAL exergame intervention for MI includes 36 training sessions with three sessions per week, each lasting around 45 minutes (30 minutes real training time) resulting in 12 weeks of training (two weeks of break/holiday allowed). The time frame and training intensity is based upon studies illustrating positive training effects in older adults performing exergame training. A training session includes an individually calculated amount of strength, cognitive-motor and balance training, which remains the same over the 12 week intervention period. Between the training sessions and exercises, rest intervals will be integrated to alleviate the acquisition of new skills. Participants are allowed to continue their usual daily business and activities during the study period. The training takes place at Physio SPArtos in Interlaken, Bern. They get well instructed on how to set up and use the system at the physio centre. The first two training sessions will be supervised one to one, after that someone will observe the training every 4 weeks to make adjustments and support the participants. The other training sessions will be done without supervision. However, there will be a physiotherapist available in case questions come up or help is needed. The compliance with the exergame training will be monitored using an attendance protocol filled in by participants.

Intervention group UI:

For the incontinent women in this study, the VITAAL exergame intervention will last over 12 weeks and consists of three parts 1) VITAAL exergame (2 sessions/week) lasting 45 minutes each (30 minutes real training time) at the physio centre, 2) PFM exercises according to a training booklet (3 sessions/week) lasting 10 minutes each at home and 3) education related to UI at home.. Between the training sessions and exercises, rest intervals will be integrated to alleviate the acquisition of new skills. Participants will be allowed to continue their usual daily business and activities during the study period. The training will take place at the physio centre SPArtos, Interlaken, Switzerland and their home. Women will get instructed on how to set up and use the system at the centre and how to do the PFM exercises at home. The VITAAL exergame training sessions will be supervised. Furthermore, every fourth week the additional weight for the strength training will be adjusted. However; the participants will be encouraged to use the system as independently as possible. The compliance with the exergame training will be monitored using an attendance protocol filled in by participants. For both groups, training compliance will be followed online by the investigators in the Web portal as each participant will have a personal login and training data will be stored in the internet-based back-end.

Control group MI:

Participants of the MI control group are instructed to do a non-individualized conventional training including 15 minutes walking exercise (in nature or on treadmill) and additional 15 minutes of strength, balance, and cognitive-motor exercises (at the therapy centre or at home). The exercises are based on recommendations from the "Beratungsstelle für Unfallverhütung" (bfu). The participants will receive a training booklet with the exercises. In total there are three different training programs which are divided according to their level of difficulty. Participants are instructed to start with the first level for four weeks and then go on to the next level for another 4 weeks. The control group training in this study includes 36 training session with three sessions per week, each lasting around 45 minutes resulting in 12 weeks of training (two weeks of break/holiday allowed). Between the training sessions and exercises, rest intervals will be integrated to alleviate the acquisition of new skills. Participants are allowed to continue their usual daily business and activities during the study period. The first training sessions take place at Physio SPArtos in Interlaken, whereas the walking can be made outside or on a treadmill. The participants get well instructed on how to do the training at the centre or at home. There will always be a supervisor at the training centre to further help and support the participants with any questions and issues. Furthermore, participants will be called every 4 weeks, to ensure social contact similar to that in the intervention group. The training components will not be individually adapted for this group. Participants in this groups will report their trainings in an attendance protocol and their additional activity in an activity protocol. In addition they need to rate the exercise intensity on each session with Borg scale.

Control group UI:

The control group training will last over 12 weeks. The training sessions will be divided in three parts 1) 30 minutes of brisk walking (2 sessions/week, 2) PFM exercises according to a training booklet (3 sessions/week) lasting 10 minutes each at home and 3) education related to UI at home. The PFM training booklet will be based on two studies that showed a reduction of incontinence in older adults while performing group pelvic floor muscle training (PFMT) and mobility exercises. The PFMT program will consist of 4 PFM exercises and will be divided into three phases allowing for the gradual progression in treatment (from first to third month), with gradual increase in difficult exercises in terms of duration, repetition and position. Each phase will last four weeks. Between the training sessions and exercises, rest intervals will be integrated to alleviate the acquisition of new skills. Participants will be allowed to continue their usual daily business and activities during the study period. The first training sessions take place at the physio centre SPArtos, Interlaken, whereas the walking can be made outside or on a treadmill. The participants get well instructed on how to do the training at home. Furthermore, participants will be called every 4 weeks, to ensure social contact similar to that in the intervention group. The training components will not be individually adapted for this group. Participants in this group will report their trainings in an attendance protocol and their additional activity in an activity protocol. The compliance with the active control intervention will be monitored using an attendance protocol filled in by participants. Furthermore, training compliance will be followed online by the investigators in the Web portal as each participant will have a personal login and training data will be stored in the internet-based back-end.

ELIGIBILITY:
Inclusion Criteria:

Both (MI & UI):

* Aged 60+ years
* Live independently, in a residency dwelling, or with care
* Standing straight for minimal 10 minutes without aids
* Visual acuity with correction sufficient to work on a TV screen
* Signed informed consent

Only MI:

- SPPB < 10 (only for the study group with MI)

Only UI:

* female
* diagnosed with mixed urinary incontinence (MUI) or urge urinary incontinence (UUI) according to the Questionnaire for Urinary Incontinence Diagnosis (QUID)
* moderate symptoms of UI (have reported at least 3 episodes of involuntary urine loss per week during the preceding 3 months)
* correct contraction of PFM must be possible
* must be able to undergo a gynaecological examination

Exclusion Criteria:

Both (MI & UI):

* Mobility impairments that don't allow to play the exergame
* Heavy noticeable cognitive impairments according to Thomman et al.
* Acute or unstable chronic diseases (e.g., recent cardiac infarction, uncontrolled high blood pressure or cardiovascular disease, uncontrolled diabetes)
* Orthopedic or neurological diseases that inhibit exergame training
* Rapidly progressive or terminal illness
* Insufficient knowledge of German
* Chronic respiratory disease
* Condition or therapy that weakens the immune system
* Cancer
* Serious obesity (BMI > 40kg/m2)

Only UI:

* Untreated chronic constipation
* Important pelvic organ prolapse
* Physiotherapy treatment or surgery for UI or pelvic organ prolapse in the past year
* Use of medications for UI or affecting skeletal muscles
* Change in hormonal replacement therapy in the last six months
* Having an active urinary or vaginal infection in the past three months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — For the Study with Urinary Incontinence only female participants will be included.
Enrollment: 40 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility assessed by recruitment rate | The recruitment rate is assessed from the beginning of September until the last participant is included in the study for approximately 2.5 months.
  The recruitment rate assesses the number of participants who were interested in participating in the study, the number of participants who signed informed consent and the number of participants who were eligible for the study.
Feasibility assessed by adherence rate | The adherence rate is assessed during the 12 week intervention period.
  The number of training sessions attended is recorded by the participants in an attendance protocol. The maximum number of training sessions during the 12-week intervention is 36 for the MI and UI groups.
Feasibility assessed by attrition rate | The attrition rate is assessed during the 12 week intervention period.
  The attrition rate is assessed by the number of participants lost during the trial. This will be recorded in an attrition protocol.
Feasibility assessed by a safety survey | The questionnaire is completed during follow-up measurements within two weeks after the intervention. The survey lasts 2 minutes.
  The study participants will receive a survey form at the end of the intervention period regarding safety during the exercises.
Feasibility assessed by a safety protocol | Safety is assessed during the 12 week intervention period.
  A protocol will be kept of all serious adverse events related to the intervention regarding safety during the exercises.
Feasibility is assessd by a survey regarding time management of the assessments | The questions will be assessed after the pre- and post-measurements within two weeks before and after the intervention. The survey lasts 1 minute.
  To investigate whether the time used for the assessments was appropriate to the study population one question will be asked about the time management of the assessments during the pre- and post-measurement and another about the time management of the assessments during the intervention. This makes it easier to assess whether the number of assessments during the study is feasible for a future study.

SECONDARY OUTCOMES:
Changes in gait speed | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The gait analysis lasts 10-15 minutes.
  Gait analysis is conducted under single- and dual-task (ST and DT) condition (UI group: with empty and full bladder) and temporal-spatial gait parameters (gait speed, step length, minimal toe clearance, cadence, stride time, swing width) are measured. Gait analysis is conducted with the Physilog. Gait speed is measured in m/s.
Changes in step length | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The gait analysis lasts 10-15 minutes.
  Gait analysis is conducted under single- and dual-task (ST and DT) condition (UI group: with empty and full bladder) and temporal-spatial gait parameters (gait speed, step length, minimal toe clearance, cadence, stride time, swing width) are measured. Gait analysis is conducted with the Physilog. Step length is measured in m.
Changes in minimal toe clearance | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The gait analysis lasts 10-15 minutes.
  Gait analysis is conducted under single- and dual-task (ST and DT) condition (UI group: with empty and full bladder) and temporal-spatial gait parameters (gait speed, step length, minimal toe clearance, cadence, stride time, swing width) are measured. Gait analysis is conducted with the Physilog. Minimal toe clearance is measured in cm. Smaller values are related to higher risk of tripping and falling. Furthermore, the coefficient of variation (CV) is calculated according to the formula CV [%] = standard deviation (SD) / mean * 100.
Changes in cadence | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The gait analysis lasts 10-15 minutes.
  Gait analysis is conducted under single- and dual-task (ST and DT) condition (UI group: with empty and full bladder) and temporal-spatial gait parameters (gait speed, step length, minimal toe clearance, cadence, stride time, swing width) are measured. Gait analysis is conducted with the Physilog. Cadence is measured in steps/min. Furthermore, the coefficient of variation (CV) is calculated according to the formula CV [%] = standard deviation (SD) / mean * 100.
Changes in stride time | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The gait analysis lasts 10-15 minutes.
  Gait analysis is conducted under single- and dual-task (ST and DT) condition (UI group: with empty and full bladder) and temporal-spatial gait parameters (gait speed, step length, minimal toe clearance, cadence, stride time, swing width) are measured. Gait analysis is conducted with the Physilog. Stride time is measured in seconds. Furthermore, the coefficient of variation (CV) is calculated according to the formula CV [%] = standard deviation (SD) / mean * 100.
Changes in swing width | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The gait analysis lasts 10-15 minutes.
  Gait analysis is conducted under single- and dual-task (ST and DT) condition (UI group: with empty and full bladder) and temporal-spatial gait parameters (gait speed, step length, toe clearance, cadence, stride time, swing width) are measured. Gait analysis is conducted with the Physilog. Swing width is measured in m.
Changes in maximal gait speed | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The gait analysis lasts 10-15 minutes.
  The maximal gait speed over at least 4 meters is measured. Gait analysis is conducted with the Physilog. Gait speed is measured in m/s.
Changes in physical performance | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The SPPB lasts 5 minutes.
  To assess physical performance the Short Physical Performance Battery (SPPB) is used resulting in a total score of 12 points with a minimum score of 0 and a maximum score of 4 for each sub-test. The SPPB consist of 3 sub-tests including a balance test (e.g. tandem stance, semi-tandem stance, single leg stance), 4-meter gait test, and 5-chair rises test. A higher score means a better balance performance.
Changes in exercise capacity | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The 1-MSTST lasts 2 minutes.
  To assess exercise capacity the 1-Minute Sit to Stand Test (1-MSTST) is used. The participants are required to rise from a chair with their arms across their chest as often as possible in one minute. The number of chair rises will be calculated.
Change in mental flexibility | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The TMT lasts 5 minutes.
  To assess mental flexibility (a part of executive functions), the Trail Making Test (TMT) is used pre- and post-intervention. This paper-pencil-test is resulting in a time value in seconds. Less time needed to conducted the test is related to better performance.
Change in interference control | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The CWIT lasts 8 minutes.
  To assess interference control (a part of executive functions), the Color Word Interference Test (CWIT) is used pre- and post-intervention. The result is a time value measured in seconds, furthermore, errors are counted. Less time and less errors is related to better performance.
Change in memory functions | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The Wechsler-Memory-Scale-Revised backwards lasts 3 minutes.
  To assess memory functions, the Wechsler-Memory-Scale-Revised backwards is used pre- and post-intervention. The test is resulting in a point score. The maximal point score is 12 points, the minimal point score is 0 points. Higher scores are related to better performance.
Changes in overall cognitive functions | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The MoCA lasts 5 minutes.
  The Montreal Cognitive Assessment (MoCA) is a test to screen several cognitive domains including memory, language, executive functions, visuospatial skills, attention, concentration, and orientation. The participants can get maximal 30 points, minimum 0 points. The MoCA can be used as a quantitative estimate of the overall cognitive abilities. A higher score indicates a higher overall cognitive function.
Changes in amount of urinary urgency (only measured in UI group) | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The USS lasts 1 minute.
  To assess the amount of urinary urgency during ST and DT walking with full bladder, the participants will complete the urinary sensation scale (USS). The USS is a 5-point likert scale developed to assess feelings of urinary urgency (i.e., intense and/or sudden need to urinate) associated with each urination. The scale goes from 1 (no urgency) to 5 (urge incontinence).
Changes in incontinence episodes (only measured in UI group) | Assessment takes place over 1 week before and after the intervention. Pre- and post-measurement changes are calculated.
  The bladder diary is a common method used to evaluate the frequency and characteristics of incontinence episodes in both research and clinical practice. The participants have to fill in a bladder diary over 7 days.
Changes in quality of life (only measured in UI group): ICIQ-UI | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The ICIQ-UI lasts 2 minutes.
  Thw International Consultation on Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI) short form is a brief and psychometrically robust patient-completed questionnaire for evaluating the frequency, severity and impact on quality of life of urinary incontinence in men and women. It is scored on a scale from 0-21. With a higher score indicating greater severity of symptoms.
Changes in pelvic floor muscle (PFM) strength (only measured in UI group) | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The PFM strength assessments lasts 10 minutes.
  The PFM strength is evaluated with 3 different assessment methods including manual muscle testing, vaginal pressure device, and electromyography (EMG).
Changes in pelvic floor muscle (PFM) endurance (only measured in UI group) | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The PFM endurance assessments lasts 5 minutes.
  The PFM endurance is evaluated with 3 different assessment methods including manual muscle testing, vaginal pressure device, and electromyography (EMG).

CONTACTS AND LOCATIONS:
Overall Officials: Eling de Bruin, Prof., Principal Investigator — ETH Zurich - Institute of Human Movement Sciences and Sport
Locations (1):
- Physio SPArtos, Bern, Interlaken, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322
- [Derived] Guimaraes V, Sousa I, de Bruin ED, Pais J, Correia MV. Minding your steps: a cross-sectional pilot study using foot-worn inertial sensors and dual-task gait analysis to assess the cognitive status of older adults with mobility limitations. BMC Geriatr. 2023 May 26;23(1):329. doi: 10.1186/s12877-023-04042-6. PMID 37237278